CLINICAL TRIAL: NCT07075159
Title: Hydrocolloid Dressings for Oculofacial Plastic and Reconstructive Wound Healing
Acronym: HCD Wound Heal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Janice Hernandez, MD (Other)
Responsible Party: Sponsor-Investigator, Janice Hernandez, MD, Instructor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 99942
Record Dates: First submitted 2025-06-23; First posted 2025-07-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wound Healing; Mohs Micrographic Surgery; Oculofacial Reconstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Wound Dressing (Experimental): At the conclusion of the surgical procedure, patients will receive topical wound dressing to surgical sutured periocular wounds
  Interventions: Device: Hydrocolloid Wound Dressing
- Antibiotic Ointment (Control) (No Intervention): At the conclusion of the surgical procedure, patients will receive topical antibiotic ophthalmic ointment to surgical sutured periocular wounds

INTERVENTIONS:
Device: Hydrocolloid Wound Dressing — one time hydrocolloid dressing application
  Other Names: DuoDERM Extra Thin dressing
  Arms: Wound Dressing

SUMMARY:
This study aims to explore the use of a hydrocolloid dressing (DuoDERM EXTRA THIN) as an alternative to the current standard of care. The dressing would be applied immediately after surgery and removed at a post-operative week 1 appointment. The dressing would eliminate the need for antibiotic ointment application and reduce the burden of post-operative care on the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* follow-up at specified intervals (1 week/6 week/3 months) in an office setting
* can give informed consent
* no patients will be excluded on the basis of gender, ethnicity, or religious background

Exclusion Criteria:

* Patients <18 years of age or >100
* allergy to pectin, gelatin, and sodium carboxymethylcellulose
* adults with impaired consent capacity
* incarcerated individuals.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with wound dehiscence | 3 months
  YES/NO type question if wound dehiscence is present after removal of the patch

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale | 3 months
  Patient and Observer Scar Assessment Scale filled out by both patient and provider at postoperative visit of both HCD Dressing and ointment. This survey is scaled from 0-10, with 0 being normal skin and 10 being very different skin. Lower scores are desired on this survey.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Hernandez, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No